CLINICAL TRIAL: NCT04904601
Title: Acute and Medium Effects of Freeze-dried Kale to go, New Superfood Supplement to Reduce Metabolic Risk in Saudi Subjects
Brief Title: Freeze-dried Kale to Reduce Metabolic Risk in Saudi Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chair for Biomarkers of Chronic Diseases (Other)
Collaborators: King AbdulAziz City for Science and Technology (Other)
Responsible Party: Principal Investigator, Dr. Dara Aldisi, Assistant Professor, Chair for Biomarkers of Chronic Diseases
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 20121503
Record Dates: First submitted 2021-04-18; First posted 2021-05-27 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Metabolic Disease
Keywords: Kale supplement; Microbiome; Obesity; Endotoxin
MeSH Terms: conditions — Obesity; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Kale (blanched freeze-dried Kale) group 1 (N=50 adult obese Saudi women)
  Placebo (Blanched Freeze-dried Peas) group 2 (N=50 adult obese Saudi women)
Who Masked: Participant, Investigator
Masking Description: Both the participant and investigator are blinded. Randomization and blinding will be done by a third party.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group: Kale (Active Comparator): This group will be given one scoop of powder of (Kale) three times a day for a total of 10g/day for 6 weeks.
  Interventions: Dietary Supplement: Kale supplement
- Placebo Group: Green Peas (Placebo Comparator): This group will be given one scoop of powder of (Green Peas) three times a day for a total of 10g/day for 6 weeks.
  Interventions: Dietary Supplement: Peas supplement

INTERVENTIONS:
Dietary Supplement: Kale supplement — Kale (blanched freeze-dried Kale) group1
  Arms: Experimental Group: Kale
Dietary Supplement: Peas supplement — placebo (Blanched Freeze-dried Peas) group2
  Arms: Placebo Group: Green Peas

SUMMARY:
Whilst obesity represents a key risk factor for the development of metabolic disease and further premature mortality, the actual type of diet may provide the 'primary insults' for inflammation affecting systemic health in the pre-diabetic state such as obesity. Specifically, previous data indicate that a high-fat diet and/or unfavorable systemic lipid profiles can impair metabolic health which may occur via inflammatory mechanisms. The study aims to conduct a randomized interventional dietary trial with Freeze-dried Kale, as a superfood, to reduce inflammation and improve lipid profile in patients with obesity. These studies will analyze the effects of this superfood on metabolic changes among obese and non-obese Saudi women. Our hypothesis is the inclusion of Brassica into the daily diet will significantly improve metabolic health, microbiota composition, lower inflammatory insults (inflammasome), and lower microbial translocation, with resulting improvements in metabolic health. The team, therefore, proposes to examine the impact of the superfood kale on lipid function (acute and medium-term) over a 4 week dietary intervention period to assess the influence on metabolic change and biomarker changes. The team intends to utilize the expertise from a broad spectrum of specialists from plant biologists, clinical and allied health care professionals, and translational scientists, to provide a unique holistic insight into the role of nutrition for metabolic health benefits in human participants. These studies will provide us with the capacity to use a directly applicable dietary supplement, freeze-dried Kale, to improve the health of people metabolically. As this is a natural product, this will have the capability to reach the market much quicker and advance research at a much faster pace. This dietary supplement will also provide an additional measure to improve the health across the general public not just those at increased risk of disease to help provide another way to improve health among Saudis.

DETAILED DESCRIPTION:
Subjects Selection:

For this study we will recruit a total of 100 obese age matched non-diabetic Saudi women, (age 18-40 years; BMI 30-40Kg/m2) through college clinics in applied medical sciences college, KSU. The study participants exclusion criteria in brief: age under 18 or above 40 years, any medical/endocrine problem that could affect energy expenditure (e.g. thyroid problems, Cushing's syndrome); chronic inflammatory disorders like rheumatoid arthritis, or long term use of steroids or other immunomodulatory like cyclosporine, azathioprine; severe depression or any psychiatric illness, claustrophobia or needle phobia.

Sample and Data Collections:

Anthropometry and body composition as well as biochemical data will be undertaken for all visits, including blood, urine and stool collection. Serum will be collected all patients for later analysis. All samples collected will be stored appropriately for biochemical analysis within the Bio-Bank facilities, in the Chair for Biomarkers of Chronic Diseases in King Saud University. All samples will be stored at -80oC following the appropriate protocol extraction methods.

Intervention:

Participants will be randomized to give either Kale (blanched freeze dried Kale) group1 or placebo (Blanched Freeze dried Peas) group2. The supplements will be given as one scoop of powder of (Kale or Green Peas) three times a day for a total of 10g/day. The follow up will be for 6 week intervention. After visit 2 will be washout period for 2 weeks, to study acute and medium effects, followed by a cross-over between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI 30-40Kg/m2 and above)
* Aged 18-40 years
* Saudi nationality
* Female

Exclusion Criteria:

* Age under 18 or above 40 years
* Any medical/endocrine problem that could affect energy expenditure (e.g. thyroid problems, Cushing's syndrome)
* Those with chronic inflammatory disorders like rheumatoid arthritis, or long term use of steroids or other immunomodulatory like cyclosporine, azathioprine; severe depression or any psychiatric illness, claustrophobia or needle phobia.
* Males
* Expatriates

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women only
Enrollment: 100 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Study the acute-term effects of freeze-dried Kale in lipid profile of obese, non-T2DM women | 2 weeks
  Differences in characteristics of total cholesterol (mmol/l), hdl-cholesterol (mmol/l), ldl-cholesterol (mmol/l) and triglycerides (mmol/l) at baseline and subsequent follow ups.
Study the medium-term effects of freeze-dried Kale in lipid profile of obese, non-T2DM women | 4 weeks
  Differences in characteristics of total cholesterol (mmol/l), hdl-cholesterol (mmol/l), ldl-cholesterol (mmol/l) and triglycerides (mmol/l) at baseline and subsequent follow ups.

SECONDARY OUTCOMES:
Study the acute and medium term effects of Kale Superfood on BMI | 6 weeks
  Differences in body mass index (BMI, kg/m2) at baseline and subsequent follow-ups
Study the acute and medium term effects of Kale Superfood on glucose levels | 6 weeks
  Differences in fasting glucose (mmol/l), at baseline and subsequent follow-ups
Study the acute and medium term effects of Kale Superfood on alanine aminotransferase levels | 6 weeks
  Differences in alanine aminotransferase (ALT, U/L)at baseline and subsequent follow-ups
Study the acute and medium term effects of Kale Superfood on aspartate aminotransferase levels | 6 weeks
  Differences in aspartate aminotransferase (AST, U/L) at baseline and subsequent follow-ups
Study the acute and medium term effects of Kale Superfood on HbA1c levels | 6 weeks
  Differences in Hemoglobin A1c (Hba1C, %), at baseline and subsequent follow-ups
Study the acute and medium term effects of Kale Superfood on insulin levels | 6 weeks
  Differences in insulin (IU/ml) at baseline and subsequent follow-ups
Study the acute and medium term effects of Kale Superfood on C-peptide levels | 6 weeks
  Differences in C-peptide levels (nmol/L) at baseline and subsequent follow-ups

CONTACTS AND LOCATIONS:
Locations (1):
- Community Health Department, Applied Medical Sciences, King Saud University, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No